CLINICAL TRIAL: NCT05499715
Title: A Phase I Clinical Study to Evaluate the Safety, the Tolerability, the Pharmacokinetic Characteristics and the Efficacy of ScTIL Injection (Genetically Modified Tumor Infiltrating Lymphocytes) in the Treatment of Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing ChineoMedical Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Aiping Zhou, Professor, Department of Medical Oncology, Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScTIL-008-2022
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Advanced Tumor of Digestive Tract or Urinary System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ScTIL injection (Experimental): In the dose escalation of the study, starting with the dose of injection of 5x10^9. If there is no DLT, followed by the second dose of 1.0x10^10 until the third dose of 2.0x10^10.
  Interventions: Biological: ScTIL injection

INTERVENTIONS:
Biological: ScTIL injection — Peripheral blood mononuclear cells (PBMCs) obtained via apheresis are used for cell preparation. PD-1 positive T cells are isolated from PBMCs, are transduced with lentivirus loaded with "enhanced receptor" and "superamplification factor", and cell number are amplified. The obtained ScTIL is used for one-time intravenous infusion.

SUMMARY:
This is an open-lable, single-arm, dose escalation and dose extension phase I clinical study of ScTIL designed to observe and evaluate the safety, the tolerance, the pharmacokinetic characteristics and the effectiveness of ScTIL in the treatment of advanced malignant solid tumors, in order to provide the basis for the future clinical research to explore the best recommended phase II dose (PR2D) and treatment scheme.

DETAILED DESCRIPTION:
This study consists of two phases: the first phase will be the dose exploration phase (Phase I), followed by the dose extension phase.

In the dose escalation of the study, 3 subjects are enrolled for 1st treatment group, starting with single dose of ScTIL injection of 5x10^9 alone. If there is no dose limiting toxicity (DLT) observed, 3 subjects are enrolled into treatment groups successively in sequential order of: Group 2: ScTIL1.0x10^10; Group 3: ScTIL 2.0x10^10.

After the completion of ScTIL reinfusion for first subject of the 1st dose group, the subject will be observed for no less than 7 days. If no serious toxic and adverse events occurres, ScTIL reinfusion for the second and third subjects will be performed. If no DLT occurres by the 21th days after completion of reinfusion for the 3rd subject, The study will proceed to the next treatment group. If 1/3 of enrolled subjects have DLT, another 3 subjects will be enrolled. In any of the dose groups, if less than 1/6 subjects have DLT, subject enrollment for the next treatment group will start. If DLT occurs in more than 2/6 of subjects, the number of subjects in the previous dose group will be reviewed. If there were only 3 subjects, 3 more subjects will be enrolled. If DLT occurs in less than 1/6 subjects, the dose will be defined as the maximum tolerable dose (MTD), and the dose escalation phase of the study will be completed. If DLT occurs in more than 2/6 subjects in the first dose group, a dose reduction exploration will be performed or the study will be terminated upon decision made by the Safety Committee.

Appropriate doses will be selected by investigator for the dose extention phase study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75, regardless of gender;
2. Eastern United States Cancer Collaborative Group (ECOG) physical condition score is 0 to1;
3. Anticipated survival > 3 months;
4. Advanced digestive tract tumor or urinary system tumor confirmed by histology or cytology;
5. Patients with unresectable locally advanced or metastatic malignant digestive or urinary system tumors who have failed at least the first-line standard treatment;
6. According to iRECIST standard, at least one tumor lesion can be measured by CT or MRI. Measurable tumor lesions are defined as the longest diameter ≥ 10mm and the scanning thickness does not exceed 5.0mm. For lymph node lesions, the short diameter ≥ 15mm;
7. PD-1 positive T cells in peripheral blood accounts for≥ 18% of total T lymphocytes (By detection standard of BD accuri C6 flow cytometer);
8. Voluntarily accept the use of peripheral blood cell apheresis to obtain cells for the preparation of ScTIL cells;
9. Sufficient bone marrow and organ functions:

   1. Hematology: neutrophils is equal to or higher than 1.5×10^9/L, platelets is equal to or higher than 75×10^9/L, hemoglobin is equal to or higher than 90g/L; total lymphocytes is equal to or higher than 60% of the lower limit of normal range;
   2. Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are both eqal to or lower than 2.5 times the upper limit of normal range (ULN) (if intrahepatic metastatic tumor exists, equal to lower than 5 times of ULN); total bilirubin (TBIL) is equal to or lower than 1.5 times of ULN;
   3. Kidney function: Creatinine (Cr) is equal to or lower than 1.5 times of ULN, or creatinine clearance is equal or higher than 60;
   4. Coagulation function: Activated partial prothrombin time (APTT) is equal to or shorter than1.5 times of ULN; international normalized ration (INR) is equal to or shorter than1.5 times of ULN;
10. Qualified patients with fertility (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence, etc.) with their partners during the trial and at least 90 days after the last medication; The blood or urine pregnancy test within 7 days before the first use of the study drug in women of childbearing age (see Appendix 8 for the definition) must be negative;
11. Study subjects must obtain informed consent to this study and voluntarily sign a written informed consent before screening for enrollment..

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence shows that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, so it is not suitable to be included in the study according to the judgment of the researcher;
2. Patients who had in recent 5 years or currently have other malignant tunors, except for cured basal cell skin cancer, in situ cervical carcinoma, and in situ lung cancer, before signing the ICF;
3. Patients who received PD-L1 monoclonal antibody treatment within 12 weeks before apheresis (including but not limited to atilizumab and dovalizumab);
4. There was active infection within 1 week before apheresis, and systemic anti-infection treatment was currently required;
5. Currently suffering from interstitial lung disease;
6. Had received immunotherapy and had ≥ grade 3 IrAE;
7. Patients with active or had autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); Except for patients with clinically stable autoimmune thyroid disease and well-controlled type I diabetes;
8. The adverse reaction of previous anti-tumor treatment has not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except for the toxicity without safety risk judged by researchers such as hair loss);
9. Received anti-tumor treatment within 2 weeks before apheresis, including but not limited to chemotherapy, radiotherapy, immunotherapy, traditional Chinese medicine with anti-tumor indications, etc., except for the following:

   1. Nitrosourea or mitomycin C within 6 weeks before harvest;
   2. Oral fluorouracils and small molecule targeted drugs were taken 1 week before apheresis.
10. Received systemic glucocorticoid (prednisone >10mg/day or equivalent dose of similar drugs) or other immunosuppressant treatment within 2 weeks before apheresis; Except for the following cases: Intermittent use of local, eye, intra-articular, intranasal and inhaled glucocorticoids; Short term use of glucocorticoids for preventive treatment (e.g. prevention of contrast agent allergy);
11. Within 4 weeks before apheresis:

    1. Have received other unlisted clinical research drugs or treatments;
    2. Having undergone major organ surgery (excluding puncture biopsy) or significant trauma, or requires scheduled hospitalization during the trial period;
    3. Used live attenuated vaccine;
12. Hepatitis B: HBsAg (+) or HBeAg (+); Or anti HBe (+)/anti HBc (+) and the DNA quantity of hepatitis B is higher than the detection limit of the research center; Hepatitis C: anti HCV positive; Treponema pallidum antibody (+);
13. Have a history of immunodeficiency, including HIV antibody test positive;
14. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular blockade, etc;
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events ≥ grade 3 occurred within 6 months before the cell reinfusion;
    3. New York Heart Association (NYHA) cardiac function rating ≥ class II or left ventricular ejection fraction (LVEF) < 50%, or structural heart disease with high risk judged by other researchers;
    4. Clinically uncontrollable hypertension;
15. Serous cavity effusion beyond clinical control as judged unsuitable for being enrolled by the researcher;
16. Known alcohol or drug dependence;
17. Mental disorders or poor compliance;
18. Pregnant or lactating women;
19. The researcher believes that the subject has a history of other serious systemic diseases or is not suitable to participate in this clinical study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 weeks after single dose of cell reinfusion
  Including cases of PR and of CR

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 12 weeks after the single dose of cell reinfusion
  The number of cases with remission and stable lesions after treatment accounted for the total number of evaluable cases
Duration of Response (DOR) | 12 weeks after single dose of cell reinfusion
  Time from complete remission (CR) or partial remission (PR) to disease progression (PD), death or last tumor evaluation
Progression-Free Survival (PFS) | 12 weeks after single dose of cell reinfusion
  From the beginning of cell therapy to the time of the first disease progression or death due to any cause
Overall survival (OS) | From single dose of cell reinfusion to death
  Time from cell reinfusion to death due to any cause
Adverse events (AEs) | 24 weeks after single dose of cell reinfusion
  According to National Cancer Institute Common Terminology Criteria for Adverse Events V5.0(CTCAE V5.0)
Detection of Lentivirus Copy Number | 12 weeks after single dose of cell reinfusion
  Dynamic changes of carrier gene copy number in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Prof. Dr., Principal Investigator — Department of oncology, Cancer hospital of Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital & Institute, Chinese Academy of Medical Sciences, Beijing, China